CLINICAL TRIAL: NCT03818958
Title: Study of the Interest of Serum Calprotectin Determination in the Diagnosis of Spondyloarthritis and to Diferenciate With Fibromyalgia
Brief Title: Seric Calprotectine in Spondyloarthritis
Acronym: Calprotect
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 17-COLL-04
Record Dates: First submitted 2019-01-21; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Spondylarthritis
MeSH Terms: conditions — Spondylarthritis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- active spondyloarthritis: subjects with active spondyloarthritis with a BASDAI greater than 4
  Interventions: Other: blood sampling
- remission spondyloarthritis: subjects presenting with a remission spondyloarthritis defined by a BASDAI less than 4
  Interventions: Other: blood sampling
- controls without spondyloarthritis: controls without spondyloarthritis or other chronic inflammatory rheumatism and without fibromyalgia
  Interventions: Other: blood sampling
- fibromyalgia: subjects with fibromyalgia
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — blood sampling

SUMMARY:
To date, there are no biomarkers in spondyloarthritis that can differentiate between spondyloarthritis and fibromyalgia or other pathologies. Fecal calprotectin is a biomarker that is increasingly used in inflammatory diseases of the digestive tract. A growing interest in this biomarker is emerging in rheumatology, several publications have focused on its interest in rheumatoid arthritis, highlighting an association between serum calprotectin levels and disease activity. In spondyloarthritis, a few studies seem to show that it could be a marker of disease activity. Although a 2012 study found no difference in serum calprotectin levels between subjects with spondyloarthritis and controls. Still others have shown that it could be a predictive factor of radiological evolution in the same disease key. These data support, despite the questionable results of the Klingberg study, the value of this dosage in spondyloarthritis. The objective of this work is to show that this assay could be useful to differentiate spondyloarthritis from other pathologies with similar clinical presentation such as fibromyalgia. Difficulties classically encountered in common practice in rheumatology.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the active line of the rheumatology department with one of the following criteria:

  * active spondyloarthritis (BASDAI >4),
  * or spondyloarthritis in low activity (BASDAI<4),
  * or fibromyalgia without associated inflammatory rheumatism,
  * or healthy subjects (without inflammatory rheumatism and without fibromyalgia.
* Patients who have not objected to the use of their samples

Exclusion Criteria:

* Minor patient
* Subject not affiliated to the social security system
* Subject deprived of liberty
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary clinic care, rheumatology patients at the CHU de NICE
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
calprotectine rate | 5 months
  blood test

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No